CLINICAL TRIAL: NCT05323487
Title: Mechanisms of Diuretic Resistance in Heart Failure
Brief Title: Mechanisms of Diuretic Resistance in Heart Failure, Aim 1
Acronym: MsDR
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: 2000032328; 1R01DK130997-01 (NIH)
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Bumetanide

STUDY DESIGN:
Intervention Model Description: This study will employ a randomized order, double-blind, repeated measures dose ranging design.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Bumetanide 10 mg (Active Comparator): Randomized to doses 10 mg, 5 mg, 2.5 mg, 1.25 mg
  Interventions: Drug: Bumetanide Injection
- Bumetanide 5 mg (Active Comparator): 5 mg Randomized to doses 10 mg, 5 mg, 2.5 mg, 1.25 mg
  Interventions: Drug: Bumetanide Injection
- Bumetanide 2.5 mg (Active Comparator): 2.5 mg Randomized to doses 10 mg, 5 mg, 2.5 mg, 1.25 mg
  Interventions: Drug: Bumetanide Injection
- Bumetanide 1.25 mg (Active Comparator): 1.25 mg Randomized to doses 10 mg, 5 mg, 2.5 mg, 1.25 mg
  Interventions: Drug: Bumetanide Injection

INTERVENTIONS:
Drug: Bumetanide Injection — Participants in balance will present to the study site Day 0 and receive their first randomized dose of bumetanide (1.25mg, 2.5mg, 5mg, or 10mg) and undergo the bio-specimen collection protocol. They will return every 3 days, allowing 2 full days washout, to receive the other doses in random sequence.

SUMMARY:
This study will employ a randomized order, double-blind, repeated measures dose ranging design. This design was chosen in order to generate multiple within-subject serial loop diuretic dose response exposures. The overall study schema will include 75 heart failure (HF) patients.

DETAILED DESCRIPTION:
The protocol will begin with pre-study determination of diuretic response at the screening visit via administration of 10 mg IV bumetanide infused over 1 hour and measuring peak Fractional Excretion of Sodium (FENa), 1-hour post completion of infusion. Participants will begin a study diet provided by the metabolic kitchen five days prior to the first study visit with randomized treatment (Day 0). Participants in balance will present to the study site Day 0 and receive their first randomized dose of bumetanide (1.25mg, 2.5mg, 5mg, or 10mg) and undergo the bio-specimen collection protocol. They will return every 3 days, allowing 2 full days washout, to receive the other doses in random sequence.

Total sodium output in response to a loop diuretic differs based on Glomerular Filtration Rate (GFR). However, a diuretic responsive participant with normal or severely reduced GFR each will achieve a similar peak FENa of approximately 20% with high dose diuretic. In a cohort of 109 hospitalized diuretic resistance (DR) HF patients that received 12.5mg bumetanide, a peak FENa <5% occurred in 66% patients. The mean FENa in this group was 2.6 ± 1.3 %, thus FENa <5% is common and a clinically relevant threshold for DR, and thus was chosen as the threshold to define diuretic resistance for the proposed study.

Participants will be asked to follow the study diet as the design seeks to decrease the variability of diuretic response introduced by variations in dietary sodium intake. For the current study, a four-gram sodium (0.8 g/kg protein) diet will be utilized. Four grams was chosen since, in prior experience, this is the average pre-study sodium intake of outpatient HF study participants and thus will facilitate rapid transition into balance.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of HF
* No plan for titration/change of heart failure medical or device therapies during the study period.
* Absence of non-elective hospitalizations in the previous 3 months.
* At optimal volume status by symptoms, exam, and dry weight
* Age > 18 years

Exclusion Criteria:

* GFR <20 ml/min/1.73m2 using the Chronic Kidney Disease- Epidemiology (CKD-EPI)equation or use of renal replacement therapies
* Use of any non-loop type diuretic in the last 14 days with the exclusion of low dose aldosterone antagonist (e.g., spironolactone or eplerenone ≤50 mg). Examples of non-loop diuretics include but may not be limited to acetazolamide (oral or IV, not ophthalmic), metolazone, Hydrochlorothiazide (HCTZ), chlorthalidone, chlorothiazide, indapamide, triamterene, amiloride, finerenone, spironolactone dose > 50mg day, eplerenone > 50mg/day,
* History of flash pulmonary edema requiring hospitalization and treatment with biphasic positive airway pressure or mechanical ventilation or a "brittle" volume sensitive HF phenotype such as an infiltrative or restrictive cardiomyopathy (i.e. amyloid cardiomyopathy, etc).
* Hemoglobin < 8 g/dL
* Pregnant or breastfeeding
* Inability to give written informed consent or comply with study protocol or follow-up visits
* Chronic Urinary retention limiting ability to perform timed urine collection procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in fractional excretion of lithium(FELi) pre-diuretic to 1-hour post IV bumetanide infusion | Baseline and 1 hour post bumetanide infusion.
  The fractional excretion of lithium is used for interrogation of sodium handling in the proximal tubule and loop of Henle. Possible values range from 0 to 100%. Change = FELi 1 hour post bumetanide infusion - FELi pre-diuretic. Different doses of bumetanide will be given at days 0, 3, 6 and 9.
Change in distal sodium reabsorption pre-diuretic to 1-hour post IV bumetanide infusion | Baseline and 1 hour post bumetanide infusion.
  The distal sodium reabsorption is used to for interrogation of how much sodium is being reabsorbed in the distal tubule. Possible values range from 0 to 100%. Distal sodium reabsorption is calculated = Fractional excretion of lithium - fractional excretion of sodium. Change in distal sodium reabsorption = distal sodium reabsorption 1 hour post bumetanide infusion - distal sodium reabsorption pre-diuretic. Different doses of bumetanide will be given at days 0, 3, 6 and 9.
Tubular diuretic efficiency at baseline | Baseline
  The tubular diuretic efficiency is used to assess the response to loop diuretics based on the amount of sodium excreted but eliminates drug delivery as source of diuretic resistance. Possible values range from 0 to 100%. Greater numbers imply better diuretic efficiency. Tubular diuretic efficiency will be compared between diuretic resistant and diuretic responsive patients using the 6 hour urine collection after bumetanide infusion.
Ratio of A to F splice variant Messenger Ribonucleic Acid (mRNA )in urinary extracellular vesicles at baseline | Baseline
  The ratio of A to F splice variant mRNA in urinary extracellular vesicles refers to the splice variants in the NKCC2 channel. The F variant has low-chloride-affinity-high-capacity, and the A variant has high-chloride-affinity-high-capacity. Possible values are greater than zero. The ratio of A to F splice variant will be compared between diuretic resistant and diuretic responsive patients. The ratio will be compared using the baseline urine sample.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Testani, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No